CLINICAL TRIAL: NCT01418586
Title: An Open Label, Randomised, Two Period, Two Treatment, Two Sequence, Crossover, Single-Dose Bioequivalence Study of Torrent Pharmaceuticals Ltd's Alfuzosin ER Tablets vs. Sanofi's Uroxatral ER Tablets in Healthy Human Subjects Under Fasted Conditions
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd's Alfuzosin ER Tablets Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Chief Investigator, Torrent Pharmaceuticals Limited
Other Study IDs: PK-06-106
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: Torrent's Alfuzosin Extended Release Tablet

SUMMARY:
Objective:

Primary objective of the present study was to assess the relative bioavailability of two formulations of Extended Release Alfuzosin 10 mg under Fasted conditions, in healthy adult male subjects after an oral administration with 7 days washout period.

Study Design:

Open-Label, Randomised, two Period, two treatment, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

(*)The volunteers were excluded from the study based on the following criteria:

* Sex: male.
* Age: 18 - 45 years. .
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

(*)The volunteers were excluded from the study based on the following criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, - - - Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd.,, Village Bhat, Gandhinagar, Gujarat, India